CLINICAL TRIAL: NCT00826670
Title: Enterobacteriaceae Producing Extended-spectrum β-lactamases (ESBL) Decolonization Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Stephen Harbarth, Médecin adjoint agrégé, Service Prévention et Contrô- le de l'Infection, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 08-161
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Enterobacteriaceae Infections
Keywords: Antibiotic resistance; ESBL carriage
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Topical decolonization (Experimental)
  Interventions: Drug: Decolonization
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Decolonization)

INTERVENTIONS:
Drug: Decolonization — Colistin sulphate (50mg 4x/d PO) + Neomycin (250mg 4x/day PO) for 10 days
  plus In the presence of urinary tract colonization choice of one of the following agents (according to susceptibility profile, creatinine clearance and individual contraindications) Nitrofurantoin (100mg 3x/day PO) or Norfloxacin (400mg 2x/day PO) for 5 days
  Arms: Topical decolonization
Drug: Placebo (Decolonization) — Placebo
  Arms: Placebo

SUMMARY:
Multidrug-resistant Enterobacteriaceae producing extended-spectrum β-lactamases (hereafter called ESBLs) have emerged as an important cause of bloodstream infection in hospitalized patients and urinary tract infections in the community. As is the case with other multidrug-resistant organisms chronic colonization is frequent, in the case of ESBLs mostly intestinal and urinary carriage.

To the investigators knowledge no randomized, placebo-controlled clinical trial has been performed to study the efficacy of a systematic ESBL eradication strategy. Eradication of ESBL carriage would cause benefits for the individual patient - by reducing the risk of infection - and for the community - by reducing transmission. Even if eradication turns out to be impossible, transient suppression of ESBL might reduce the likelihood of transmission and thus still be beneficial from an ecologic perspective.

The purpose of the proposed study is to test the hypothesis that the administration of a 10 day course of oral antibiotics active against ESBLs can lead to decolonization of ESBL carriage in hospitalized patients.

ELIGIBILITY:
Inclusion Criteria:

Patients can be enrolled into the study provided that all of the following criteria are met:

1. Microbiologically documented rectal carriage of ESBL-producing Enterobacteriaceae, without signs and symptoms of active infection with ESBL-producing Enterobacteriaceae at any body site
2. Patient must give written informed consent to participate in the study. The informed consent can be given by the legal representative if necessary.

Exclusion Criteria:

1. Women who are pregnant or nursing
2. Active infection
3. Treatment with antimicrobial agents with activity against ESBL-producing Enterobacteriaceae
4. Contraindication to the use of one of the study drugs (e.g. renal insufficiency with creatinine clearance < 30 ml/min)
5. Patient already enrolled in another study, or in the present study for a previous episode
6. Psychiatric disorder or unable to understand or to follow the protocol directions
7. Permanent indwelling urinary catheter that can not be changed
8. Resistance of the ESBL-producing Enterobacteriaceae to one of the study drugs
9. Known hypersensitivity to one of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Rate of eradication of carriage with ESBL-producing Enterobacteriaceae at day 28 post-treatment | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva Universits Hospitals, Geneva, Switzerland

REFERENCES:
- [Derived] Huttner B, Haustein T, Uckay I, Renzi G, Stewardson A, Schaerrer D, Agostinho A, Andremont A, Schrenzel J, Pittet D, Harbarth S. Decolonization of intestinal carriage of extended-spectrum beta-lactamase-producing Enterobacteriaceae with oral colistin and neomycin: a randomized, double-blind, placebo-controlled trial. J Antimicrob Chemother. 2013 Oct;68(10):2375-82. doi: 10.1093/jac/dkt174. Epub 2013 May 29. PMID 23719234